CLINICAL TRIAL: NCT05696730
Title: Holistic Wellbeing in COPD: The Communication About Sexuality (COSY) Randomized Controlled Trial
Brief Title: Holistic Wellbeing in COPD: Communication About Sexuality (COSY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Anja Frei, Principal Investigator, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COSY
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Chronic Disease; Lung Diseases, Obstructive; Respiratory Disease
Keywords: Quality of life; COPD; Intimacy and sexuality; Communication intervention; Physical activity; Randomized controlled trial
MeSH Terms: conditions — Chronic Disease; Lung Diseases, Obstructive; Respiration Disorders; Pulmonary Disease, Chronic Obstructive; Sexuality; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the control or intervention group.
Who Masked: Investigator
Masking Description: Due to the kind of intervention and the organizational structure of the study centre, neither patients nor assessors can be blinded, but data analysts will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication intervention about sexuality in people with COPD (Experimental): Communication intervention. Individual counselling to improve holistic well-being by addressing sexuality and to increase adherence for long-term physical activity given the correlation with sexual activity.
  Interventions: Other: Communication intervention about sexuality in people with COPD
- 30 minutes counselling and intervention material per request after the RCT (No Intervention): Usual care. Participants will have the possibility to receive a brief version of the intervention on request (30 minutes counselling and intervention material) at the end of the 3-months follow-up assessment visit.

INTERVENTIONS:
Other: Communication intervention about sexuality in people with COPD — COSY is a communication intervention which consists of one face to face counselling (75 min) and two 30-min telephone call counselling.
  Patients assigned to the intervention group will get the COSY communication intervention with a special focus on the positive impact of sexuality on wellbeing plus specific motivation for physical activity. Together with the patient, a personalized re-enforcement instrument, the COSY-Compass, is elaborated to set individual goals and motivation for physical activity over the whole intervention period (3 months).
  Participants will learn to understand the positive effect of regular physical activity on physical, mental, and cognitive wellbeing and a more fulfilling sex life as well as get inspiration about the spectrum and possible expressions and manifestations of caring and intimacy with oneself.
  Arms: Communication intervention about sexuality in people with COPD

SUMMARY:
The aim of this study is to assess the effectiveness of a communication intervention about sexuality on quality of life and other outcomes like physical activity, exercise capacity and health status in people with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Human sexuality is a universal part of living and associated with quality of life and mental and physical health benefits. Improved sexual relationships and sexual activity might also be an intrinsic motivator to stay physically active. However, problems with sexuality and loss of sexual drive are common in older and chronically ill people like persons with chronic obstructive pulmonary disease (COPD). In persons with COPD sexuality is rarely addressed during medical consultations and the topic is not sufficiently researched despite the fact that a thorough assessment of quality of life is incomplete without considering sexuality.

Based on this background, the investigators developed an instrument that supports healthcare professionals to start and shape communication about sexuality: COSY. The COSY intervention consists of four tools (communication leaflet for health care professionals, application guidance, pictorial representation of the spectrum of intimacy for health care professionals, patient information booklet) and aims to sensitize persons with COPD with the topic sexuality.

The aim of this study is to assess the effectiveness of the COSY communication intervention on quality of life and other outcomes like physical activity, exercise capacity and health status in people with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Diagnosis of COPD, defined as forced expiratory volume in 1s/forced vital capacity (FEV1/FVC)<70% predicted, FEV1<80 % predicted after bronchodilation corresponding to a Global initiative on Obstructive Lung Disease (GOLD) stage II-IV
* Knowledge of German language to understand study material and assessments and being able to give informed consent as documented by signature

Exclusion Criteria:

* Unstable COPD at the time of recruitment, unstable cardiovascular comorbidities, severe depression, or predicted life expectancy of less than one year, as judged by the referring clinician or the intervention physician

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Quality of life in old age (CASP-12) | Change from baseline to 3 months
  The CASP is a validated measure developed specifically to assess quality of life in old age by the total score of the CASP-12 (Control, Autonomy, Self-realization and Pleasure) german short-version of the CASP-19 scale; 12 questions; 4-point Likert-type-scale ranging from 1 (never) to 4 (often)

SECONDARY OUTCOMES:
Physical activity (PROactive physical activity in COPD instrument, clinical visit version [C-PPAC]; domains amount and difficulty) | Change from baseline to 3 months, measured during 1 week
  The C-PPAC is a validated and reliable hybrid tool combining a short patient-reported outcome questionnaire and two activity monitor variables (assessed by the accelerometer ActiGraph®) to measure physical activity in COPD patients in the two domains amount and difficulty; 12 questions; 5-point Likert-type-scale (item scores 0-4, scale 0-100, higher socres indicating higher amonunt of/less difficulty with physical activity)
Functional exercise capacity (1-min Sit-to-Stand [STS] test) | Change from baseline to 3 months
  The 1-min STS test assesses the number of repetitions that the patient completes the full sit-to-stand movement from a standard chair (i.e. standing up from a chair and sitting down again) during one minute
COPD-specific health-related quality of life (Chronic Respiratory Questionnaires [CRQ] Subscales) | Change from baseline to 3 months
  The CRQ is a validated tool to assess COPD-specific health-related quality of life with four domains: Dyspnea, fatigue, emotional function, mastery domain. The total CRQ contains 20 questions responded to on a 7-point Likert-type scale, ranging from 1 to 7 with lower scores indicating worse HRQoL
COPD-specific health status / Symptoms (COPD Assessment Test; CAT) | Change from baseline to 3 months
  The CAT measures the impact of COPD on a person's health status, covering the most burdensome symptoms and limitations of COPD; 8 questions; 6-point Likert-type scale (item scores: 0-5, overall score 0-40 with higher score indicating poorer health status)
Health status (Feeling Thermometer; FT) | Change from baseline to 3 months
  The FT is a visual analogue scale for overall health state ranging from 0 (worst health you can imagine) to 100 (best healthy you can imagine)
Exacerbations of COPD (event based, patient reported) | At 3-months follow-up assessment visit
  The event-based definition required an increase in symptoms and an increase in dosage of or new prescription of systemic corticosteroids and/or antibiotics
Symptoms of anxiety and depression (Hospital Anxiety and Depression Scale; HADS) | Change from baseline to 3 months
  The HADS assesses symptoms of anxiety and depression and contains 14 questions responded to on a 4-point Likert-type scale ranging from 0 to 3 with higher scores indicating a higher symptom score

OTHER OUTCOMES:
Experience and feedback with the counselling program of the health professionals | At 3-months follow-up assessment visit
  Semi-structured interview, outcomes will be qualitatively assessed (no scale is used)
Experience and satisfaction with the counselling program of the participants | At 3-months follow-up assessment visit
  Semi-structured interview, outcomes will be qualitatively assessed (no scale is used)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Frei, PhD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich / Epidemiology, Biostatistics and Prevention Institute, Zurich, Switzerland